CLINICAL TRIAL: NCT05667792
Title: Examination of the Effects of Video-Based Games on Balance, Trunk Proprioception, Motivation and Quality of Life in Individuals With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, İlkan Cicek, Postgraduate, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MustafaKU-PTIlkan
Record Dates: First submitted 2022-08-01; First posted 2022-12-29 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: CP (Cerebral Palsy)
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Study Group- 4-11 age (Experimental)
  Interventions: Device: Microsoft Kinect 360; Other: Pediatric Rehabilitation
- Control Group-4-11 age (Placebo Comparator)
  Interventions: Other: Pediatric Rehabilitation
- Study Group- 12-18 age (Experimental)
  Interventions: Device: Microsoft Kinect 360; Other: Pediatric Rehabilitation
- Control Group-12-18 age (Placebo Comparator)
  Interventions: Other: Pediatric Rehabilitation

INTERVENTIONS:
Device: Microsoft Kinect 360 — Balance and trunk proprioception games will be selected and played for the children to be included in the treatment. Children will play these games with their own body movements.
  Arms: Study Group- 12-18 age; Study Group- 4-11 age
Other: Pediatric Rehabilitation — Bobath therapy

SUMMARY:
In the study we planned, 42 individuals diagnosed with cerebral palsy will be divided into 2 groups according to age groups. Individuals aged 4-11 will be included in the child group, and individuals aged 12-18 will be included in the adolescent group. Individuals with cerebral palsy in the child and adolescent group will also be randomized and divided into treatment and control groups. In addition to the conventional treatment created in accordance with neurodevelopmental treatment approaches, video-based virtual reality games will be played for a total of 10 weeks for treatment groups in both age groups. The patients will be followed up with a video-based game application for an average of 20 minutes, after the physiotherapy and rehabilitation application, which consists of an average of 45 minutes, twice a week. Individuals in the control group in both age groups will be followed for 10 weeks with conventional treatment created in accordance with neurodevelopmental treatment approaches.

The entire sample will be evaluated at the beginning of the study and at the end of the 10th week. Our main aim in the study is to compare the effects of video-based games applied in different age groups on balance, trunk proprioception, motivation and quality of life.

DETAILED DESCRIPTION:
A total of 42 patients with cerebral palsy who agreed to participate in the study, 22 patients between the ages of 4-11 and 22 patients between the ages of 12-18, will be included. Parents of the patients will be informed about the study.

42 individuals diagnosed with cerebral palsy will be divided into 2 groups according to age groups. Individuals aged 4-11 will be included in the child group, and individuals aged 12-18 will be included in the adolescent group. Individuals with cerebral palsy in the child and adolescent group will also be randomized within themselves and divided into treatment and control groups. In addition to conventional treatment created in accordance with neurodevelopmental treatment approaches, video-based virtual reality games will be played for a total of 10 weeks for treatment groups in both age groups. The patients will be followed up with an average of 20 minutes of video-based games, after the physiotherapy and rehabilitation application, consisting of an average of 45 minutes, twice a week. Individuals in the control group in both age groups will be followed for 10 weeks with conventional treatment created in accordance with neurodevelopmental treatment approaches.

A treatment plan will be created for the entire sample group according to neurodevelopmental treatment approaches. In the content of the treatment plan; In order to regulate muscle tone and increase sensory input, intramuscular stretching and soft tissue mobilization, exercises that improve protective, balance and correction reactions, and support the development of postural control will be included. In addition, studies aimed at ensuring proper posture and increasing body awareness during standing without support, facilitation of trunk extension will be carried out. For the development of postural control in the same position, facilitation of trunk elongation and weight transfer to the affected and less affected side will be emphasized. Exercises will be performed on stepping and descending from the affected and less-affected side. Supported with appropriate hand grips, forward jumping with two feet, one foot, and weight transfer on one foot will be carried out.

In the evaluation of the patient, the pediatric motivation scale, balance, trunk proprioceptive sense and quality of life will be evaluated at the 1st and 10th weeks.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with spastic type CP with bilateral and unilateral involvement Volunteer to participate in the study Be between the ages of 4-18 Being at 1/2 level according to Gross Motor Function Classification System Cooperate with assessments Cooperating with virtual reality therapy

Exclusion Criteria:

* Botulinum toxin administration in the last 6 months Having had any surgical operation in the last 6 months

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
One Leg Standing Test | beginning and week 10
  The one-leg stance test is a test in which the time to stand on balance is measured on the right and left extremities of the patient, and evaluates the static balance. Change will be evaluated.
Caliper Clinometer | beginning and week 10
  Caliper inclinometer is a phone protractor application used to measure angle changes in the relevant region. In the evaluation of trunk proprioception, the person is in a sitting position with the back unsupported and the feet not touching the ground, while the arms are positioned crossed on the trunk. Change will be evaluated
Pediatric Motivation Scale | beginning and week 10
  The scale consists of 21 items divided into 6 subsections (effort-importance, interest-pleasure, competence, relationship, autonomy, value-benefit) and enables the evaluation of the child's motivation towards the rehabilitation program from her own perspective.The total score is 119. The higher the score, the higher the motivation. Change will be evaluated.
Pediatric quality of life questionere pedsQL for Children | beginning and week 10
  The Children's Quality of Life Scale was developed to measure the quality of life of children and adolescents aged 2-18.It is scored between 0-100, with the highest score being 100. Change will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Hatay Mustafa Kemal Üniversitesi, Antakya, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No